CLINICAL TRIAL: NCT05990946
Title: A Prospective, Randomized, Controlled Study to Evaluate the Impact of Remote Symptom Management Via Smartphone App Based on Electronic Patient-Reported Outcomes on Rehabilitation Exercise Adherence After Minimally Invasive Surgery in Lung Cancer Patients
Brief Title: Smartphone-based Remote Symptom Monitoring to Improve Postoperative Rehabilitation Exercise Adherence After Video-assisted Thoracic Surgery (VATS) for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Xiaojuan Yang, Nurse Practitioner, Zhongshan People's Hospital, Guangdong, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K2022-285
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Lung Neoplasms, Non-Small Cell Lung Cancer; Postoperative Complications; Patient Reported Outcome Measures; Telerehabilitation; Exercise Therapy
Keywords: Exercise Adherence; ePRO; Remote Monitoring; Postoperative Rehabilitation; Symptom Management
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will complete ePRO symptom severity scores on the PSA-Lung questionnaire via the smartphone app on discharge and post-discharge days 3, 7, 14, 21, 28. Alerts are triggered if any of 5 core symptoms scored ≥4, prompting remote clinician feedback and guidance on symptom management.
  Interventions: Device: ePRO based Remote Symptom Management provide by a mobile phone app
- Control Group (No Intervention): Participants randomized to the control group will complete ePRO symptom severity scores on the PSA-Lung questionnaire via the smartphone app on discharge and post-discharge days 3, 7, 14, 21, 28, without clinician alerts.

INTERVENTIONS:
Device: ePRO based Remote Symptom Management provide by a mobile phone app — Alerts are triggered if any of 5 core symptoms scored ≥4, prompting remote clinician feedback and guidance on symptom management. This is facilitated through the "Shuyu" mobile application, which serves as the platform for monitoring symptoms and communication.
  Other Names: mobile phone app for Remote Symptom Management
  Arms: Intervention Group

SUMMARY:
Brief Summary: This randomized controlled trial aims to evaluate whether active remote symptom monitoring and management via a smartphone app utilizing electronic patient-reported outcomes (ePRO) can improve adherence to prescribed outpatient pulmonary rehabilitation exercises among postsurgical lung cancer patients. Eligible patients will use the app for perioperative care and be randomized to an intervention group receiving ePRO-based symptom monitoring with clinician feedback or a control group receiving ePRO without feedback. The primary outcome is rehabilitation exercise adherence rate over 1 month after discharge. If proven effective, the app-enabled remote rehabilitation model can be scaled up to enhance recovery for more postoperative patients.

Due to slower-than-expected recruitment, an interim analysis was introduced through a protocol amendment. The amendment was approved by the Ethics Committee before conducting the analysis, and the plan was incorporated into the updated study record. The interim review evaluated feasibility and informed the addition of mean weekly exercise duration as a co-primary endpoint with adjusted statistical thresholds.

DETAILED DESCRIPTION:
Adherence to postoperative pulmonary rehabilitation exercises is crucial but challenging to address in lung cancer patients after hospital discharge. Pain, fatigue, cough and other symptoms may hinder adherence. This study will enroll 224 patients undergoing Video-assisted thoracic surgery (VATS) for lung Cancer. All patients will use a smartphone app for perioperative care and periodic PRO measurement. Before discharge, patients will be randomized 1:1 to an intervention group or control group. The intervention group will complete ePRO symptom severity scores on the PSA-Lung Scale questionnaire on discharge and post-discharge days 3, 7, 14, 21, 28. Alerts are triggered if any of 5 core symptoms scored ≥4, prompting remote clinician feedback and guidance. The control group will complete ePRO without clinician alerts. The primary outcome is rehabilitation exercise adherence rate over 1 month after discharge. Secondary outcomes include postoperative complications, hospital readmissions, symptom changes, exercise participation rate, and patient satisfaction. If proven effective, this innovative rehabilitation model can be scaled up to enhance recovery for more postoperative patients.

Due to slower-than-expected recruitment, the study protocol was amended to introduce one interim analysis. The protocol amendment was reviewed and approved by the Ethics Committee before the analysis was conducted. The interim analysis was performed using aggregated, de-identified data by an independent monitoring group, without disclosing any individual-level unblinded outcomes to investigators. Based on the interim findings, mean weekly exercise duration was added as a co-primary endpoint alongside 1-month adherence. Statistical thresholds for interim testing were adjusted using an O'Brien-Fleming alpha-spending approach (interim p < 0.006).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Undergoing minimally invasive lung cancer resection
* Able to use smartphones and complete electronic questionnaires
* Signed informed consent

Exclusion Criteria:

* conversions to open thoracotomy during surgery
* ECOG score > 1
* Received neoadjuvant therapy
* Previous lung resection surgery
* Unable to exercise due to physical limitations
* Continuous systemic corticosteroid use within 1 month before enrollment
* Unresolved toxicity above Grade 1 from previous treatments
* Significant comorbidities or medical history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation exercise adherence rate over 1 month after discharge | From the day of discharge to 30 days after discharge
  Rehabilitation exercise adherence rate over 1 month after discharge, defined as the proportion of patients completing the prescribed outpatient exercise regimen.
Mean weekly exercise duration over 1 month after discharge | From discharge to 30 days after discharge.
  Mean weekly exercise duration measured over the first 30 days post-discharge. This endpoint was added following a protocol amendment and interim review. Interim testing used an O'Brien-Fleming alpha-spending boundary.

SECONDARY OUTCOMES:
Post-discharge pulmonary complication rate | From the day of discharge to 30 days after discharge
30-day hospital readmission rate | From the day of discharge to 30 days after discharge
Changes in symptom severity scores from discharge to 30 days | From the day of discharge to 30 days after discharge
Patient satisfaction scores | From the day of discharge to 30 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- No.2 Sunwen East Rd., Zhongshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Not available. The individual participant data collected in this study will not be shared with external researchers.

REFERENCES:
- [Derived] Yang X, Zhang Q, Ye C, Cheng Y, Wu J, Liang Y, Su J. Factors Influencing Symptom Severity at Discharge after Lobectomy and Sublobar Resection Through Video-assisted Thoracoscopic Surgery. Interdiscip Cardiovasc Thorac Surg. 2025 Aug 5;40(8):ivaf170. doi: 10.1093/icvts/ivaf170. PMID 40811025
- [Derived] Su J, Ye C, Zhang Q, Liang Y, Wu J, Liang G, Cheng Y, Yang X. Impact of Remote Symptom Management on Exercise Adherence After Video-Assisted Thoracic Surgery for Lung Cancer in a Tertiary Hospital in China: Protocol for a Prospective Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 1;14:e60420. doi: 10.2196/60420. PMID 39610048